CLINICAL TRIAL: NCT04451486
Title: A Phase I Study to Evaluate The Use of Autologous-Derived Adult Peripheral Small Blood Stem Cells to Enhance Osseointegration of Guided Bone Regeneration in Implant Surgery
Brief Title: A Phase I Study of SB Cell for the Enhanced Osseointegration of Guided Bone Regeneration in Implant Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N201709009
Record Dates: First submitted 2020-06-15; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Guided Bone Regeneration
Keywords: SB cell、autologous、Osseointegration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment dose 1 (Experimental): 1x10*5 CD61-Lin- cells /0.25mL DPBS
  Interventions: Drug: SB cells
- Treatment dose 2 (Experimental): 1x10*6 CD61-Lin- cells /0.25mL DPBS
  Interventions: Drug: SB cells
- Treatment dose 3 (Experimental): 1x10*7 CD61-Lin- cells /0.25mL DPBS
  Interventions: Drug: SB cells

INTERVENTIONS:
Drug: SB cells — 1x10*5 CD61-Lin- cells /0.25mL DPBS
  Arms: Treatment dose 1
Drug: SB cells — 1x10*6 CD61-Lin- cells /0.25mL DPBS
  Arms: Treatment dose 2
Drug: SB cells — 1x10*7 CD61-Lin- cells /0.25mL DPBS
  Arms: Treatment dose 3

SUMMARY:
This is a Phase 1 study to evaluate the safety profile of autologous-derived SB cells to enhance osseointegration of GBR in patients undergoing dental implant surgery.

DETAILED DESCRIPTION:
This is a Phase 1 study to evaluate the safety profile of autologous-derived SB cells to enhance osseointegration of GBR in patients undergoing dental implant surgery.

Enrolled subjects eligible to receive GBR procedure will be sequentially assigned to 1 of 3 treatment cohorts as follows:

Treatment dose 1 group：1×10*5 CD61-Lin- cells /0.25mL DPBS Treatment dose 2 group：1×10*6 CD61-Lin- cells /0.25mL DPBS Treatment dose 3 group：1×10*7 CD61-Lin- cells /0.25mL DPBS

After receiving the autologous SB cells solution mixed with 1 mL bone substitute, each first treated subject at each cohort will be followed up to 4-weeks. After the first subject at each cohort (3 subjects) complete a 4-weeks follow-up period, if investigator and sponsor judge that there is not either a safety concern or a dose-limiting toxicity (DLT) criteria is not met, 2 additional subjects within each cohort will be enrolled. A Data Safety Monitoring Committee will be conveyed after the first 3 treated subjects at each cohort complete undergo the dental implant procedure (12-weeks follow-up after GBR) to evaluate the safety and preliminary efficacy of SB cells administered during a GBR procedure, and will provide recommendations regarding study modification, continuation to enroll next subject(s), cohorts or study termination.

If the committee recommends further subject enrollment, sequential recruitment will continue until subjects for each treatment cohort are enrolled, treated and followed up to 24-weeks after GBR (12-weeks after dental implant) unless there is a safety concern judged by investigator, sponsor, or a dose-limiting toxicity (DLT) criteria is met. Once this situation occurs, the committee will assess the progress and safety data of all subjects enrolled, and will provide recommendations regarding study modification, continuation to enroll next subject in that or other cohorts, or will recommend study termination.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 20 years old and over;
2. Sign of informed consent form;
3. Patients with one missing tooth with D2, D3 bone density;
4. Gums environment defined as alveolar bone height of 10 mm and above, bone width 8 mm and above;
5. Have only one missing maxillary or mandibular posterior tooth (No. 4, 5, 6 or 7) who require a GBR prior to a dental implant.
6. Bone defect(s) must be present with at least two walls missing.
7. The opposing dentition must be nature teeth or fixed crowns or bridges on natural teeth or implants. Removable prostheses or dentures opposing the study implants are not allowed;
8. Subject is able to understand and comply with protocol requirements, instructions and protocol stated restrictions

Exclusion Criteria:

1. Patients who have inadequate organ function described as below:

   1. ANC < 1.5 x 109/L
   2. Platelets < 100 x 109/L
   3. Hb < 9 g/dL
   4. Serum bilirubin < 1.5 x the upper limit of normal (ULN)
   5. Aspartate aminotransferase (AST [SGOT]) < 2.5 × the ULN
   6. Alanine aminotransferase (ALT [SGPT]) > 2.5 × the ULN
   7. Serum creatinine > 1.5 mg/dL or a measured creatinine clearance < 60 mL/min;
2. History of neoplastic disease and had been treated with chemotherapy;
3. Uncontrolled Diabetes Mellitus;
4. Dialysis patients;
5. Patients with cardiovascular disease;
6. Osteoporosis patients and patients taking bisphosphonates;
7. History of radiation therapy to the head and neck;
8. Patients with temporomandibular disorder;
9. Pregnant or nursing women;
10. Presence of conditions requiring chronic routine prophylactic use of antibiotics (history of rheumatic heart disease, bacterial endocarditis, cardiac valvular anomalies, prosthetic joint replacements);
11. Medical conditions requiring prolonged use of steroids;
12. Physical handicaps that would interfere with the ability to perform adequate oral hygiene;
13. Use of any investigational drug or device within the 30-day period immediately prior to implant surgery on study day 0;
14. Alcoholism or drug abuse;
15. Patients infected with HIV;
16. Current smokers, ;
17. Local inflammation, including untreated periodontitis;
18. Mucosal diseases such as erosive lichen planus;
19. History of local radiation therapy;
20. Presence of osseous lesions;
21. Unhealed extraction sites;
22. Persistent intraoral infection;
23. Patients with inadequate oral hygiene or unmotivated for adequate home care;
24. Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability.
25. Patient with a pathology present near the site of dental implantation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2021-04-25 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | Throughout the study, an average of 1 year

SECONDARY OUTCOMES:
The maximum tolerated dose (MTD) of autologous-derived Small Blood Stem Cells in patients undergoing dental implant surgery. | Throughout the study, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Schneider R. Prosthetic concerns about atrophic alveolar ridges. Postgrad Dent. 1999;6(2):3-7. PMID 11360322
- [Background] de Baat C, Kalk W, van 't Hof M. Factors connected with alveolar bone resorption among institutionalized elderly people. Community Dent Oral Epidemiol. 1993 Oct;21(5):317-20. doi: 10.1111/j.1600-0528.1993.tb00783.x. PMID 8222609
- [Derived] Feng SW, Su YH, Lin YK, Wu YC, Huang YH, Yang FH, Chiang HJ, Yen Y, Wang PD. Small blood stem cells for enhancing early osseointegration formation on dental implants: a human phase I safety study. Stem Cell Res Ther. 2021 Jul 2;12(1):380. doi: 10.1186/s13287-021-02461-z. PMID 34215319